CLINICAL TRIAL: NCT03150823
Title: Effects of Ascending and Descending Direct Current on Grip Strength. Evaluation Through Dynamometry and Myofeedback. Randomized, Controlled Trial.
Brief Title: Effects of Ascending and Descending Direct Current on the Handgrip Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Principal Investigator and Clinical Professor, Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6031205
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Muscle Strength
Keywords: Direct current; Galvanic current; Handgrip Force; Palmar Grip; Dynamometry; Miofeedback

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upward Direct Current (Ascending Effect) (Experimental): Group subjected to a direct current application (Longitudinal Galvanization) in which the anode is placed at the distal level and the cathode at the proximal level. This would be an excitatory effect of the nervous system.
  Interventions: Procedure: Upward Direct Current (Ascending Effect)
- Downward Direct Current (Descending Effect) (Experimental): Group subjected to a direct current application (Longitudinal Galvanization) in which the cathode is placed at the distal level and the anode at the proximal level. This would be an inhibitory effect of the nervous system.
  Interventions: Procedure: Downward Direct Current (Descending Effect)
- Sham Direct Current (Sham Comparator): Group to which an electrical installation will be carried out without emission of part of the electrotherapy equipment. The electrodes will be applied longitudinally to the participants with the equipment switched off.
  Interventions: Procedure: Sham Direct Current

INTERVENTIONS:
Procedure: Upward Direct Current (Ascending Effect) — Application of direct current (Galvanic) in milliamperes current which varies according to the positioning of the electrodes. In the ascending stream direct current (Ascending effect) the proximal cathode and distal anode are placed, a excitatory effect on the nervous system being described in theory.
  Arms: Upward Direct Current (Ascending Effect)
Procedure: Downward Direct Current (Descending Effect) — Application of direct current (Galvanic) in milliamperes current which varies according to the positioning of the electrodes. In the descending stream direct current (Descending effect) the proximal anode and distal cathode are placed, a sedative and analgesic effect on the nervous system being described in theory.
  Arms: Downward Direct Current (Descending Effect)
Procedure: Sham Direct Current — Installation of electrotherapy equipment off (Sham tratment).
  Arms: Sham Direct Current

SUMMARY:
Electrical stimulation currently has a wide range of clinical applications, being used for activities such as strengthening, pain control, edema management, or inflammation control after injury or surgery. One of the classic forms of electrotherapy is the Direct current (galvanic current), which stands out for its unique effects (polar and interpolar effects) and that are not achieved with other modalities of electrotherapy. Within these effects those activators or suppressors of nervous system activity are described. One of the applications of direct current is to produce sedation or excitation on the nervous system through longitudinal applications (longitudinal galvanization). This application technique is known as the upstream or downstream effect of the direct current or "Leduc Effect", in which it is postulated that an ascending type longitudinal galvanization has excitation effects of the central and / or peripheral nervous system. The study will evaluate the influence of the upward and downward direct current effect when performing a manual dynamometer test while monitoring by miofeedback in college students.

DETAILED DESCRIPTION:
Methodological Design

1. Type of research: Experimental study, of type randomized clinical trial (RCT).
2. Conceptual definition of the variables;

   * Ascending effect: Excitation effect on the nervous system by a longitudinal direct current application (Longitudinal Galvanization), in which the anode is placed at the distal level and the cathode at the cranial level.
   * Descending effect: Sedative effect on the nervous system by a longitudinal direct current application (Longitudinal Galvanization), in which the anode is placed at the cranial level and the cathode at the distal level.
   * Placebo: Phenomenon by which a patient's symptoms can be improved by treatment with a safe substance, ie a substance with no effects directly related to the treatment of symptoms or illness (a placebo will be applied in a control group).
3. Operational definition of variables;

   * Maximum Handgrip strength: Maximum Strength in kilograms evaluated through manual dynamometry test the time for a grip. Force values are recorded in an Excel table displaying data in kilograms evaluated. (Manual hydraulic dynamometer brand JAMAR® be used).
   * Maximum activation threshold: measured in microvolts (μV) by a miofeedback device on the muscular belly of the dominant forearm in the flexopronator muscles. The GYMNA® electrotherapy equipment model MYO 200 were used.
   * Direct upnstream current (Ascending Effect): it were applied through an electric direct current quantified in milliamps (mA) in a longitudinal galvanizing technique with the catode electrode in proximal position. The GYMNA® electrotherapy equipment model COMBI 500 were used.
   * Direct downstream current (Descending effect): it were applied through an electric direct current quantified in milliamps (mA) in a longitudinal galvanizing technique with the anode electrode in proximal position. The GYMNA® electrotherapy equipment model COMBI 500 were used.
   * Placebo: was applied through a circuit switched off (sham intervention). The GYMNA® electrotherapy equipment model COMBI 500 were used.
4. Definition of the type of variable;

   * Maximum Handgrip strength: dependent, quantitative, reason variable.
   * Maximum activation threshold: dependent variable, quantitative, reason variable.
   * Direct upstream current (Ascending effect): independent variable, qualitative, nominal variable.
   * Direct downstream current (Descending effect): independent variable, qualitative, nominal variable.
   * Placebo: independent variable, qualitative, nominal variable.
5. Place of research;

   The study will be conducted in the laboratory of Physiotherapy Rehabilitation Science Faculty, building C5, 401 room floor, Campus Casona de la Universidad Andrés Bello, Av. Fernández Concha 700, Las Condes.
6. Methodology;

   This research has the characteristics of an experimental randomized design. The study will be carried out in the physiotherapy laboratory, room 401, 4th floor, building C5 of the Andrés Bello University (UNAB), faculty of rehabilitation sciences, Casona Campus, Las Condes commune, Calle Fernández Concha Nº700, Santiago de Chile.

   The sample was selected from the university population that is part of the Faculty of Rehabilitation Sciences (FCR) of the Andrés Bello University Andrés. The study will be presented to the ethics committee of the Metropolitan Health Service East (SSMO). Once the study is approved by the committee, the investigation will begin. The study group will be determined through a simple random sampling process using a random number table (RAND Corporation random number table ). The sample will be recruited from a survey with closed questions built according to the proposed inclusive and exclusive criteria, which will allow the selection of participants according to the proposed icriteria at work. The number of participants for the research will be taken for convenience. As inclusion criteria the following have been established; Participants over 18 years of age, people who do not show discomfort or pain when performing manual grasping with the dominant limb, and students belonging to the Faculty of Rehabilitation Sciences (FCR). As exclusion criteria were considered: people with musculoskeletal pathologies of hand, wrist and elbow in the last 6 months, osteosynthesis or prosthesis materials in areas of current application, peripheral neurological pathologies such as neuropraxis or nerve cuts, alterations of sensibility such as hypoesthesia, anesthesia or hyperesthesia, alterations in the skin of the areas of application of the current and monitoring through miofeedback that include burns, wounds, scars, apprehension or fear of the application of electrotherapy, and non-completion of the evaluation protocol / intervention designed for the study or abandonment of the same.

   Three stages of conducting for this study were designated. The first stage called "Sampling Stage" will be 3 weeks long. This stage consisted of the application of the survey to the target population and its subsequent analysis based on the information collected, allowing a first filter selection of the potential participants. The survey will be applied to the students of the FCR of the Universidad Andrés Bello. The first filter will be given by the questions of the survey itself. Participants who meet the proposed participation requirements will then be physically contacted and invited to participate in the study. Interested students will be given a detailed explanation of the project and will be asked, in case they wish to participate, to give their consent in writing. Informed consent reflects the 4 principles of bioethics in order to safeguard the integrity of the person.

   The second stage of the design was called "Evaluation Stage" had a duration of 2 weeks. In this stage will be evaluate the ability to perform manual grip in a dynamometry test will following the protocol established in the research. The test was performed in a scenario with the same working conditions of the study. In addition, it was explained at this stage everything concerning the characteristics of electrical stimulation used and evaluation procedure through myofeedback device, as well as its form of application according to the proposed intervention protocol. Stage two marked a second filter to discard the participants who presented discomfort, or problems to execute the manual grip by dynamometry. Once this stage is completed, the final number of participants will be included in the study (sample), which will allow to advance to stage 3 or "Experimentation Stage". This stage will last for 5 weeks. The sample will be randomized to establish 3 working groups, group 1 or "Upstream direct current group," group 2 or "Downstream direct current group", and a third or "control group". Randomization will be performed by the director of the, through a simple random sampling process using a number table (RAND Corporation number tables), thus reducing possible selection bias. After this process a definitive list of participants will be counted by group and that only the director of the study will handle. Demographic variables (secondary variables) for each group, including age, body mass index (BMI) and gender, will be tabulated, in addition to the primary variables such as "Maximum handgrip strength" (Kilograms) and "Maximum electromyographic surface activation threshold "(Microvolts) measured with dynamometry and miofeedback respectively in a first evaluation before the application of electrotherapy or" Pre-intervention Evaluation". This allowed to determine the initial characteristics for each group to establish possible initial comparisons and to finalize the measurements once having the results. An evaluator 2 will record the "Maximum Handgrip Force" of the dominant limb of each individual while at the same time that through the miofeedback (MF) procedure the "Electromyographic Activation Threshold". The maximum grip strength will be evaluated following the research protocol. Evaluator 2 will request three executions within 15 seconds, leaving a rest interval of 60 seconds between each attempt (according to the proposed protocol based on the work of Watanabe et al.). The records of the primary variables in this stage will be defined as "Maximum pre-intervention handgrip force" (PRE MHF) and "Maximum electromyographic activation threshold of pre-intervention surface" (PRE MEAT). The evaluator 2 will tabulate the values of the three executions handgrip attempts with their corresponding electromyographic values in an Excel® worksheet highlighting the best value of grip strength (maximum grip force) which will be recorded as the maximum handgrip pre intervation value. Following the process of evaluation of grip strength, the director will refer each participant to the corresponding intervention group, ie "Direct Upstreamcurrent" group, "Direct Downstream current" or "Control" group, according to the randomization of the sample. In the laboratory there will be three working boxes, one for each intervention procedure. In the laboratorywere three physical therapist, one by box and one for each procedure. The therapist will not know the values obtained from the evaluations of force or electromyographic activation threshold performed by the evaluator 2, nor will they be aware of the participants that will make up the other study groups. Interveners will be familiar with the application of direct current modality, since they will be kinesiologists with more than 3 years of experience. Each controller will work using the GYMNA® COMBI 500 equipment. In the application will work with a single channel of the equipment in each individual, applying one of the electrodes inside a bucket with water at a temperature of 25 °C. The participant must introduce the hand of the dominant upper extremity into the bucket, while the other electrode will close the circuit in the ventral region of the forearm thus generating a longitudinal galvanizing arrangement. For Group 1 the red electrode will be used distally in the bucket, and the black electrode in the forearm area (direct current). On the other hand, in Group 2 the black electrode in the bucket and the red electrode in the forearm (downward direct current) will be used, while for the control group the electrode will be used either red or black distally and the other in The forearm, because the difference will be that the first two groups will be applied a current of 4mA, based on safety recommendations when applying this type of currents (theoretical framework), while the control group will not receive stimulation. None of the three groups will experience any sensation, because with the programmed currents current densities are imperceptible. With these parameters a current density of 0.02mA / cm2 is obtained, considering that it will work with rectangular carbon rubber electrodes of 48cm2 area. To ensure that the installation is skewed, the studio director will mask the color of the channel electrodes (red and black) by means of a white insulation tape, so that the differences between the colors of the electrodes will not be distinguished, thus ignoring Is the positive or negative. Only the letter A or B will appear on the label. The application time for each group will be 12 minutes, according to the electrotherapy application protocol established for the investigation, which generated a current dose of 48mA / min according to the work intensity indicated previously. Participants of the three groups will be installed in wooden chairs in a sedentary position. The electrotherapy equipment will be placed on the side of the dominant limb with its screen facing towards the participant's feet so that the adjusted intensity value is not displayed. After completion of the current application time, the participant will leave the intervention laboratory and the evaluation room will be conducted, where the dynamometry test was applied. The holding force will be recorded again following the measurement protocol, recording again 3 attempts, respecting the same interval times performed before the application of direct current. The evaluator 2 will record in a Microsoft Excel® worksheet, the Kilograms of the best maximum grip strength of the 3 trials and their corresponding value in μV of the electromyographic surface register. These values will be defined as "Maximum post-intervention handgrip force" (POST MHF) and "Maximum electromyographic activation threshold of post-intervention surface" (POST MEAT).

   After completing the weeks prepared for the measurement, 1 month will be left for the data ordering and analysis of the information. This task will be taken be the study director who will be responsible for storing and ordering the data received by the evaluators and intervenors. For this process the Microsoft Excel® program will be used. The descriptive statistics for the primary variables "Maximum Handgrip force Difference" (DIF MHF), "Maximum Pre-intervention Handrgrip force" (PRE MHF) and "Maximum Post-Intervention Handgrip force" (POST MHF) will use as analysis measures, averages, fashion, frequencies and standard deviation. For the variables "Maximum electromiographic activation threshold difference" (DIF MEAT), "pre-intervention electromyographic activation threshold" (PRE MEAT) and "post-intervention electromyographic activation threshold" (POST MEAT), the averages, frequencies and standard deviation between and within groups will be recorded. This information will also be presented in the form of bar charts. The secondary variables including age and bone mass index will be expressed as averages, while sex will be expressed as frequency. In terms of inferential statistics, SHAPIRO WILK (S-WILK) normality test will be used to determine if the distribution of data obtained for the primary and secondary variables is normal or not, and according to this will select the statistical test of greater relevance , ANOVA test if the data distribute normal or Mann Whitney test if the data do not distribute normal. For the statistical calculation, the SPSS v.24.0 program will be used. Once the statistical analysis is done, a period of 1 month will be considered for the analysis of the results, discussion and results.
7. Measurement protocol of Dynamometric Handgrip strenght and of Miofeedback. The measurement of grip strength will be carried out in the physiotherapy laboratory, room 401, 4th floor, building C5 of Andrés Bello University (UNAB), FCR, Casona Campus, Las Condes Commune, Avenida Fernández Concha No. 700, Santiago , Chile. Initially participants are instructed to sit in a straight back chair with dimensions of 42cm high, 46cm wide by 40cm long, 10º tilt back and dimensions of 43cm high by 46cm wide. Each participant should be located with; Feet supported flat on the floor, trunk erected in contact with the back, head and neck in neutral position, adducted shoulder, in neutral rotation, elbow flexed in 90º, forearm in prono neutral supination, without any surface support and wrist in position Neutral test.67 The test will use a Jamar® hydraulic hand-held dynamometer, weighing 600gr and whose dimensions are 26cm long and 13cm wide. The instrument allows double reading on a measurement scale of up to 200lbs / 90kg. For the investigation the Kilograms will be considered as a measurement value. In addition it has five levels of manual adjustment, being fixed in the second level. The evaluator will install 2 (active) electrodes on the anterior region of the forearm in order to evaluate the "Maximum Activation threshold with surface electromyography" by the miofeedback device. The electrodes shall be placed 3cm from the mid-point of elbow flexion following the axis from that point to the middle finger. A third electrode (reference electrode) will be installed at the midpoint of the brachial biceps muscle following a line between the anterior portion of the acromion and the midpoint of the elbow flexion fold. The estimated time of measurement per participant is 10 minutes considering time of explanation of the test and the execution itself.

   The grip strength will be evaluated in 3 opportunities. Participants will be instructed to position themselves correctly in the work station and apply maximum force for 3 seconds, requesting the maximum effort in each attempt, turning the dynamometer marker to 0lbs / kg after each grip. The rest between measurements will be 60 seconds81. Subsequently, the best measured value of the 3 trials performed and its corresponding value obtained with the MF were recorded. An Excel® spreadsheet was used to record data for pre-application of electrotherapy.
8. Application of electrotherapy protocol. The intervention will be carried out in the physiotherapy laboratory, room 401, 4th floor, building C5 of Andres Bello University (UNAB), faculty of rehabilitation sciences, Casona Campus, Las Condes commune, Calle Fernández Concha Nº700, Santiago , Chile. After the force measurement, the participants will be placed in the electrotherapy station, where each person was placed in a chair (Annex 9). The subject should support the trunk at the back of the chair at a 90 ° angle of hip flexion, knee and both feet resting on the floor, the distal end of the dominant upper limb inserted into a plastic bucket with water at 25 ° C. For the application of electrotherapy, the Combi 500 brand Gymna® will be used.

Two carbon electrodes of 7.5cm long and 6cm wide were also covered by damp conducting pads 9,5cm long and 8cm wide, resulting in an area of 48cm2. One of the electrodes will be placed inside the bucket with water while the other will be fixed to the proximal third of the forearm on its anterior face (Annex 9), closing the circuit with a longitudinal galvanization. For group 1 (direct current) the red electrode will be used distally in the bucket with water, and the black electrode in the area of the forearm. For group 2 (direct downward current) the black electrode in the bucket and the red electrode in the forearm will be applied, while for group 3 (control) the electrode will be used interchangeably, either red or black distally and the other in the forearm. The controllers will ignore the sign of each electrode, because they will be masked with a white tape with only numbers A or B. The director of the study will only know the polarity of the electrode and it will be the one who will indicate if it is the electrode A or B that will In the bucket. In groups 1 and 2 direct current will be applied at 4mA for 12 minutes (dose 48mA.min). The control group did not apply any intensity keeping the equipment on but no emission during the same time as groups 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Students of the Faculty of Rehabilitation Sciences.
* Participants older than 18 years of age.
* Participants who do not show discomfort or pain when performing manual grip in the dominant hand.

Exclusion Criteria:

* Musculoskeletal pathologies of hand, wrist or elbow in the last 6 months.
* Materials of osteosynthesis or prosthesis in areas of application.
* Peripheral neurological pathologies such as or nerve compression cuts.
* Sensitivity alterations such as hypoesthesia, anesthesia or hyperesthesia in the upper limbs.
* Alterations in the skin of the application areas, such as burns, wounds, scars.
* Apprehension or fear of the application of electrotherapy.
* Non-completion of the evaluation / intervention protocol, designed for the study or abandonment of the same.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Difference of Maximum handgrip force | Baseline and 1 hours later (1 session of treatment), assessed as up to 1 month.
  Comparing maximum handgrip strength pre and post application of upward and downward direct current intervention
Difference of Maximum Electromiographic Activation Threshold | Baseline and 1 hours later (1 session of treatment), assessed as up to 1 month.
  Comparing maximum Electromiographic Activation pre and post application of upward and downward direct current intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Andrés A de la Barra Ortiz, Mg., Principal Investigator — Study Principal Investigator
Locations (1):
- Universidad Andrés Bello, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michelle H. Cameron, Physical Agents in Rehabilitations 2003, Elsevier. Cap. VIII, P, 220.
- [Background] Rodríguez Martin JM, Galvanismo V. En J. Rodríguez, Electroterapia en fisioterapia. 2 Edición. Madrid: Editorial Médica Panamericana, 2004.
- [Background] Avendaño Coy, A. Ferri Morales, E. Sánchez Sobrados, A. Ceciaga Ajuria. Efectos de la galvanización sobre el umbral excitomotor. Estudio sobre individuos sanos. Rev Iberoam Fisioter Kinesiol 2001;4(1):00-00.
- [Background] Kahn J. Iontophoresis. Phys Ther. 1984 Jun;64(6):956, 959. doi: 10.1093/ptj/64.6.956a. No abstract available. PMID 6728918
- [Background] Raiman J, Koljonen M, Huikko K, Kostiainen R, Hirvonen J. Delivery and stability of LHRH and Nafarelin in human skin: the effect of constant/pulsed iontophoresis. Eur J Pharm Sci. 2004 Feb;21(2-3):371-7. doi: 10.1016/j.ejps.2003.11.003. PMID 14757511
- [Background] Guy RH, Delgado-Charro MB, Kalia YN. Iontophoretic transport across the skin. Skin Pharmacol Appl Skin Physiol. 2001;14 Suppl 1:35-40. doi: 10.1159/000056388. PMID 11509905
- [Background] Galvani, L. Opere edite ed inedite del Professore Luigi Galvani raccolte e pubblicate dall'Accademia delle Science dell'Istituto di Bologna. Bologna: Dall'Olmo; 1841.
- [Background] Panus PC, Ferslew KE, Tober-Meyer B, Kao RL. Ketoprofen tissue permeation in swine following cathodic iontophoresis. Phys Ther. 1999 Jan;79(1):40-9. PMID 9920190
- [Background] Kalia YN, Naik A, Garrison J, Guy RH. Iontophoretic drug delivery. Adv Drug Deliv Rev. 2004 Mar 27;56(5):619-58. doi: 10.1016/j.addr.2003.10.026. PMID 15019750
- [Background] Fujita M, Hukuda S, Doida Y. The effect of constant direct electrical current on intrinsic healing in the flexor tendon in vitro. An ultrastructural study of differing attitudes in epitenon cells and tenocytes. J Hand Surg Br. 1992 Feb;17(1):94-8. doi: 10.1016/0266-7681(92)90021-s. PMID 1640154
- [Background] Conjeevaram R, Banga AK, Zhang L. Electrically modulated transdermal delivery of fentanyl. Pharm Res. 2002 Apr;19(4):440-4. doi: 10.1023/a:1015135426838. PMID 12033377
- [Background] Oh SY, Guy RH. Effects of iontophoresis on electrical properties of human skin in vivo. Int J Pharmacol 1995;124:137-42.
- [Background] Watanabe T, Owashi K, Kanauchi Y, Mura N, Takahara M, Ogino T. The short-term reliability of grip strength measurement and the effects of posture and grip span. J Hand Surg Am. 2005 May;30(3):603-9. doi: 10.1016/j.jhsa.2004.12.007. PMID 15925174
- [Background] O'Driscoll SW, Horii E, Ness R, Cahalan TD, Richards RR, An KN. The relationship between wrist position, grasp size, and grip strength. J Hand Surg Am. 1992 Jan;17(1):169-77. doi: 10.1016/0363-5023(92)90136-d. PMID 1538102
- [Background] Innes E. Handgrip strength testing: A review of the literature. Aust Occup Ther J 1999; 46(3):120-140.)
- [Background] Mathiowetz V, Kashman N, Volland G, Weber K, Dowe M, Rogers S. Grip and pinch strength: normative data for adults. Arch Phys Med Rehabil. 1985 Feb;66(2):69-74. PMID 3970660
- [Background] Kozin SH, Porter S, Clark P, Thoder JJ. The contribution of the intrinsic muscles to grip and pinch strength. J Hand Surg Am. 1999 Jan;24(1):64-72. doi: 10.1053/jhsu.1999.jhsu24a0064. PMID 10048518
- [Background] Glass JM, Stephen RL, Jacobson SC. The quantity and distribution of radiolabeled dexamethasone delivered to tissue by iontophoresis. Int J Dermatol. 1980 Nov;19(9):519-25. doi: 10.1111/j.1365-4362.1980.tb00380.x. PMID 7429701
- [Background] Margin del Socorro Martínez Matheus, Principios de Electroestimulación y terminología Electroterapéutica Primea edición Bogotá año 2006 P, 34 a 39.
- [Background] McNeal DR: 2000 years of electrical stimulation. In: Hambrecht FT Ryswick JB, eds: Functional Electrical Stimulation: Applications Neural Prostheses, New York, 1977 Marcel Dekker.
- [Background] Volta, A. Le opere di Alessandro Volta (edizione nazionale), I vol. Milano; Hoepli; 1918.